CLINICAL TRIAL: NCT01534754
Title: Mesalazine and/or Lactobacillus Casei in Maintaining Remission of Symptomatic Uncomplicated Diverticular Disease of the Colon: a Double-blind, Double-dummy, Placebo-controlled Study
Brief Title: Mesalazine and/or Lactobacillus Casei in the Diverticular Disease of the Colon
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Cristo Re (Other)
Responsible Party: Principal Investigator, Giovanni Brandimarte, MD; PhD, Hospital Cristo Re
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-00064322-25
Record Dates: First submitted 2012-02-04; First posted 2012-02-17 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Diverticular Disease of the Colon
MeSH Terms: interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mesalazine (Active Comparator): Active mesalazine 800 mg, 2 tablets/day for 10 days/month plus Lactobacillus casei placebo, 1 sachet/day for 10 days/month.
  Interventions: Drug: Mesalazine 800 mg
- Lactobacillus casei (Active Comparator): Active Lactobacillus casei, 1 sachet/day for 10 days/month plus mesalazine 800 mg placebo, 2 tablets/day for 10 days/month.
  Interventions: Drug: Lactobacillus casei
- Mesalazine plus Lactobacillus casei (Active Comparator): Active mesalazine 800 mg, 2 tablets/day plus active Lactobacillus casi, 1 sachet/day for 10 days/month.
  Interventions: Drug: Mesalazine plus Lactobacillus casei
- Placebo (Placebo Comparator): Mesalazine 800 mg placebo, 2 tablets/day and Lactobacillus casei placebo, 1 sachet/day for 10 days/month.
  Interventions: Drug: Mesalazine placebo plus Lactobacillus casei placebo

INTERVENTIONS:
Drug: Mesalazine plus Lactobacillus casei — Active Mesalazine 800 mg, 2 tablets/day and active Lactobacillus casei, 1 sachet/day for 10 days/month for one year.
  Arms: Mesalazine plus Lactobacillus casei
Drug: Mesalazine placebo plus Lactobacillus casei placebo — Mesalazine 800 mg placebo, 2 tablets/day and Lactobacillus casei placebo, 1 sachet/day for 10 days/month for oe year.
  Arms: Placebo
Drug: Mesalazine 800 mg — Active mesalazine 800 mg, 2 tablets/day and Lactobacillus casei placebo, 1 sachet/day for 10 days/month for one year.
  Arms: Mesalazine
Drug: Lactobacillus casei — Mesalazine 800 mg placebo, 2 tablets/day and active Lactobacillus casei, 1 sachet/day for 10 days/month for one year.
  Arms: Lactobacillus casei

SUMMARY:
This is a multi-centre, randomised, double blind, double-dummy, parallel groups, placebo-controlled trial was conducted in a population of patients suffering from symptomatic uncomplicated diverticular disease in order to investigate which is the best treatment in preventing relapses of the disease.

Patients were randomly divided in double-blind fashion in one of the following groups:

Group A. Active mesalazine 800 mg, 2 tablets/day for 10 days/month plus Lactobacillus casei placebo, 1 sachet/day for 10 days/month;

Group B. Active Lactobacillus casei, 1 sachet/day for 10 days/month plus mesalazine 800 placebo, 2 tablets/day for 10 days/month;

Group C. Active mesalazine 800 ng, 2 tablets/day plus Active Lactobacillus casei, 1 sachet/day for 10 days/month;

Group D. Mesalazine 800 mg placebo, 2 tablets/day and Lactobacillus casei placebo, 1 sachet/day for 10 days/month.

The main objective was to assess the safety and the efficacy of mesalazine and/or Lactobacillus casei in maintaining remission of symptomatic uncomplicated diverticular disease

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of diverticular disease diagnosed for the first time or established by previous colonoscopy
* symptomatic episode of uncomplicated diverticular disease no more than 4 weeks prior to study entry
* patients who have given their free and informed consent.

Exclusion Criteria:

* acute diverticulitis (both complicated and uncomplicated)
* diverticular colitis
* active or recent peptic ulcer
* chronic renal insufficiency
* allergy to salicylates
* patients with intended or ascertained pregnancy, lactation
* women of childbearing age not using contraceptives
* lactulose-lactitol use in the two weeks before the enrolment and during the study
* presence of diverticulitis complications (fistulas, abscesses, and/or stenoses)
* use of probiotic preparations either prescribed or over-the counter within two weeks prior to study entry
* inability to give a valid informed consent or to properly follow the protocol
* patients with active malignancy of any type, or history of a malignancy (patients with a history of other malignancies that have been surgically removed and who have no evidence of recurrence for at least five years before study enrolment were also acceptable)
* recent history or suspicion of alcohol abuse or drug addiction
* any severe pathology that can interfere with the treatment or the clinical or instrumental tests of the trial
* use of NSAIDS for one week before and throughout the study period (only paracetamol was permitted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of patients maintaining remission of symptomatic uncomplicated diverticular disease of the colon | one year

SECONDARY OUTCOMES:
Safety of the treatments | one year
  Number of participants with adverse events
Influence of severity of diverticulosis on number of patients maintaining remission of symptomatic diverticular disease of the colon | one year
Concomitant diseases | one year
  Influence of concomitant diseases on remission maintenance

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Brandimarte, M.D., Principal Investigator — Head of Gastroenterology, Hospital "Cristo Re" - Rome
Locations (14):
- Italy (14):
  - Hospital Bonomo, Andria, Bari
  - Hospital Policlinico, Bari, Bari
  - Hospital "Pulgiese-Ciaccio", Catanzaro, Catanzaro
  - Hospital "Padre Pio", Vasto, Chieti
  - Hospital "Ospedali Riuniti", Foggia, Foggia
  - Hospital "S. Maria Goretti", Latina, Latina
  - Hospital "Humanitas", Rozzano, Milano
  - Ospedale Civile Hospital, Popoli, Pescara
  - Hopsitla Policlinico, Reggio Calabria, Reggio Calabria
  - Hospital "S. Giuseppe", Albano Laziale, Rome
  - Hospital "G.B. Grassi", Ostia Antica, Rome
  - Hospital "S. Eugenio", Rome, Rome
  - Hospital "P. Colombo", Velletri, Rome
  - Hospital "Cristo Re", Rome

REFERENCES:
- [Derived] Tursi A, Brandimarte G, Elisei W, Picchio M, Forti G, Pianese G, Rodino S, D'Amico T, Sacca N, Portincasa P, Capezzuto E, Lattanzio R, Spadaccini A, Fiorella S, Polimeni F, Polimeni N, Stoppino V, Stoppino G, Giorgetti GM, Aiello F, Danese S. Randomised clinical trial: mesalazine and/or probiotics in maintaining remission of symptomatic uncomplicated diverticular disease--a double-blind, randomised, placebo-controlled study. Aliment Pharmacol Ther. 2013 Oct;38(7):741-51. doi: 10.1111/apt.12463. Epub 2013 Aug 19. PMID 23957734